CLINICAL TRIAL: NCT06656221
Title: A Prospective, Single-Center Study Evaluating the Efficacy and Safety of Glofitamab Combined With Orelabrutinib and Bortezomib in Patients With High-Risk Mantle Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Prof., Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Glo-MCL
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — obinutuzumab; glofitamab; Bortezomib; orelabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glofitamab-Orelabrutinib-Bortezomib (Experimental): Participants will receive 2000 mg of obinutuzumab on Days 1-2 of Cycle 1, 2.5 mg of glofitamab on Day 8 of Cycle 1, 10 mg of glofitamab on Day 15 of Cycle 1, followed by 30 mg of glofitamab on Day 1 of Cycles 2-12.
  Participants will receive 1.6 mg/m² of bortezomib on Days 1, 8, and 15 of Cycles 1-12.
  Participants will receive 150 mg/day of orelabrutinib on Days 1-21of Cycles 1-12.
  The duration of one cycle is 21 days.
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab; Drug: Bortezomib; Drug: Orelabrutinib

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab pre-treatment is given intravenously at a dose of 2000mg on Cycle 1 Days 1-2
Drug: Glofitamab — Glofitamab is given intravenously at a dose of 2.5mg on Cycle 1 Day 8. Glofitamab is given intravenously at a dose of 10mg on Cycle 1 Day 15. Glofitamab is given intravenously at a dose of 30mg on Day 1 of Cycles 2-6
Drug: Bortezomib — Bortezomib is given intravenously at a dose of 1.6 mg/m² on Days 1, 8, and 15 of Cycles 1-12.
Drug: Orelabrutinib — Orelabrutinib is given orally at a dose of 150 mg daily on Days 1-21 of Cycles 1-12.

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of Glofitamab combined with Orelabrutinib and Bortezomib in patients with high-risk mantle cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥ 18 years at the time of signing Informed Consent Form and willingness to comply with study protocol procedures
* Participants with MCL
* Meets any of the following high-risk criteria: blastoid/pleomorphic morphology; high Ki-67 (≥ 30%); TP53 aberration; del(17p); complex karyotype; MIPI score ≥ 6.2; early progression after first-line treatment (<24 months); presence of other high-risk genetic mutations (KMT2D, NSD2, NOTCH1, CDKN2A, NOTCH2, SMARCA4, CCND1)
* Life expectancy ≥ 12 weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1, or 2
* At least one bi-dimensionally measurable (≥ 1.5 cm) nodal lesion, or one bi-dimensionally measurable (≥ 1 cm) extranodal lesion, as measured on CT scan
* No bone marrow involvement: ANC ≥ 1.0 × 10^9/L; bone marrow involvement: ANC ≥ 0.5 × 10^9/L
* No bone marrow involvement: PLT ≥ 75 × 10^9/L; bone marrow involvement: PLT ≥ 25 × 10^9/L
* No bone marrow involvement: Hgb ≥ 8 g/dL; bone marrow involvement: Hgb ≥ 7 g/dL
* Adequate renal function, defined as measured or estimated creatinine clearance ≥ 30 mL/min

Exclusion Criteria:

* Contraindication to any of the individual components of Glofit-Orela-Borte
* Known active infection at the time of enrollment
* Positive test results for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HBsAg] serology): Patients with occult or prior HBV infection (defined as negative HbsAg and positive hepatitis B core antibody [HbcAb]) may be included if HBV DNA is undetectable, provided that they are willing to undergo DNA testing on Day 1 of every cycle and every three months for at least 12 months after the last cycle of study treatment and appropriate antiviral therapy
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing): Patients who are positive for HCV antibody are eligible only if PCR is negative for HCV RNA
* History of other malignancies that could affect compliance with the protocol or interpretation of results
* Active autoimmune disease requiring treatment
* Primary or secondary CNS lymphoma at the time of recruitment
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | Up to 2 years
  CR rate, defined as the proportion of patients with a best overall response of CR at any time during the study, as determined by the investigator using 2014 Lugano Response Criteria

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  ORR, defined as the proportion of patients with a best overall response of CR or PR at any time during the study, as determined by the investigator using 2014 Lugano Response Criteria.
Duration of Response (DoR) | Up to 2 years
  DoR, defined as the time from the first occurrence of a documented objective response (PR or CR) to disease progression or death from any cause (whichever occurs first) according to the 2014 Lugano Response Criteria, as determined by the investigator.
Duration of Complete Response (DoCR) | Up to 2 years
  DoCR, defined as the time from the first occurrence of a documented CR to disease progression or death from any cause (whichever occurs first) according to the 2014 Lugano Response Criteria, as determined by the investigator.
Progression-Free Survival (PFS) | Up to 2 years
  PFS, defined as the time from the first study treatment to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator using 2014 Lugano Response Criteria.
Overall Survival (OS) | Up to 2 years
  OS, defined as the time from the first study treatment to the date of death from any cause.
Incidence and severity of adverse events | Up to 2 years
  Incidence and severity of adverse events, with severity determined according to the NCI CTCAE v5.0 grading scale, except CRS that shall be graded using ASTCT CRS grading criteria 2019

IPD SHARING:
Plan to Share IPD: No